CLINICAL TRIAL: NCT06702319
Title: İzmir Democracy University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation
Brief Title: Effects of Externally Focused Shoulder Stabilization Exercises on Individuals With Rotator Cuff Tendinopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Collaborators: Buca Seyfi Demirsoy State Hospital (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXTERNALFOCUS
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Pain; Rotator Cuff Tendinitis
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home exercise program (No Intervention): A total of at least 23 Participants will receive the home exercise program for 6 weeks.
- internal focus exercise program (Experimental): A total of at least 23 Participants will receive the internal focus exercise program for 6 weeks.
  Interventions: Other: Exercise
- external focus exercise program (Experimental): A total of at least 23 Participants will receive the external focus exercise program for 6 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Home exercises and home exercises with internal focus exercises or external focus exercises
  Arms: external focus exercise program; internal focus exercise program

SUMMARY:
This study aims to evaluate the effectiveness of externally focused shoulder stabilization exercises on range of motion, pain, handgrip strength, and proprioception in patients with rotator cuff tendinopathy. For the study, 69 patients will be randomly divided into three groups: Home Program Group (HPG), Internal Focused Exercise Group (IFEG), and External Focused Exercise Group (EFEG). The treatment period for all three groups will be 6 weeks. Shoulder range of motion, pain, handgrip strength, joint position sense, and shoulder function (WORC and QuickDASH) of the three groups will be evaluated at baseline and after intervention. IFEG will do the exercises with a physiotherapist twice a week. During the exercise, the patient will be allowed to focus on the body parts while performing the movement. EFEG will do the exercises with a physiotherapist twice a week. The patient will be allowed to focus on a point outside the body, namely the effect of the movement, during the exercise. In the management of HPG patients will be provided with an exercise brochure. At the conclusion of the study, the three groups will be compared and evaluated using appropriate statistical analyses to assess the outcomes and determine any significant differences between them.

DETAILED DESCRIPTION:
Rotator Cuff Tendinopathy Treatment Various strategies are used in the treatment of rotator cuff tendinopathy as conservative, mini-invasive, and surgical treatments. Conservative treatment includes rest, non-steroidal anti-inflammatory drugs, steroid injections, and physiotherapy methods (Chaudhury et al. 2010). The primary goal in physiotherapy applications is the restoration of normal shoulder movement patterns. It focuses on eliminating the loss of flexibility, movement, and strength that cause pain and regaining functions (Kibler, 2003). The response of tendon cells to load depends on both frequency and load. Tendon cells seem to be programmed to perceive a certain level of stress. Adequate doses of mechanical loading provide repair in the tendon. On the other hand, inadequate stimulation can prevent or slow down healing (Arnocky et al. 2007, Camargo et al. 2014).

Focus of attention Focus of attention refers to the place where a person pays attention while performing a certain movement. Wulf et al. (1998) conducted the first study on the focus of attention. When a person focuses on body parts while performing a movement, it is called internal focus, and when a person focuses on something outside the body, that is, the effect of the movement, it is called external focus. Studies show that external focus is effective in balance, performance, and motor learning (Park et al., 2015; Wulf et al., 2016). It has been determined that external focus is effective in improving motor learning and function (Castillo-Vejar et al., 2022). It has been observed that performing exercises with an external focus provides a decrease in the degree of perceived exertion (Lohse et al., 2011). In a study, the effects of internal focus, external focus, and the application without focus conditions on balance performance were evaluated. As a result, a positive effect of external focus on balance was found. Internal focus has been reported to cause a loss of performance on balance compared to the control group (Wulf et al., 2003).

This study aims to determine whether there is a difference between home exercise program, internal focus exercise, and external focus exercise in patients with Rotator Cuff Tendinopathy.

Exercise Programs Initially, patients will receive training (30 minutes) to ensure that the exercises are applied correctly and to encourage patient compliance.

Home program group (HPG): In addition to medical treatment, a home exercise program with a brochure will be given to the home exercise group. The exercise program includes; posture exercises, codman exercises, wand exercises, strengthening exercises in all directions of the shoulder, and wall ball rolling exercises. It will be stated that they will do the exercises regularly and follow the given recommendations and come for a check-up at the end of 6 weeks. During this period, individuals will be contacted by phone and interim follow-ups will be made.

Internal Focused Exercise Group (IFEG): A home program will also be given to this group. In addition, participants will do the exercises with a physiotherapist twice a week. The exercises will be applied in the physiotherapy unit of Buca Seyfi Demirsoy Hospital. In this group, internal focus will be used during the exercise. During the exercise, the patient will be allowed to focus on the body parts while performing the movement. For example; while doing the ball rolling exercise on the wall, "While applying pressure to the ball on the wall with your hand, draw a circle clockwise." The exercise program includes; posture exercises, codman exercise, wand exercises, strengthening exercises in all directions of the shoulder, and ball rolling exercises on the wall.

External Focused Exercise Group (EFEG): The home program will also be given to this group. In addition, participants will do the exercises with a physiotherapist twice a week. The exercises will be applied in the physiotherapy unit of Buca Seyfi Demirsoy Hospital. In this group, external focus will be used audibly and visually during the exercise. The patient will be allowed to focus on a point outside the body, namely the effect of the movement, during the exercise. For example; while drawing a circle on the wall and rolling a ball on the wall, giving the command "Draw a circle by applying pressure to the ball on the wall, staying inside the circle." and using audible external focus such as counting the number of movements and giving directions during the exercise. The exercise program includes; posture exercises, codman exercises, wand exercises, strengthening exercises in all directions of the shoulder, and rolling a ball on the wall exercises.

Statistical method(s) The normal distribution of the obtained data will be examined and the method will be determined according to the distribution. The differences before and after the application in one group and after the training between the three groups will be examined. The results will be interpreted and discussed by comparing them with the literature. At the end of the study, statistical analyses will be performed using the SPSS 26.0 program. The conformity of all variables to normal distribution will be investigated using visual (histogram and probability graphs) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). Descriptive analyses will be given using the number and percentage (%) values for categorical variables, median and interquartile range (IQR) for variables that are not normally distributed, and mean and standard deviation (x±ss) for variables that are normally distributed. One-way variance analysis and post hoc tukey analysis will be performed in the comparison of variables that are normally distributed. In the comparison of data that are not normally distributed, the Kruskal Wallis test and one-way ANOVA test for post hoc statistics will be performed to determine the groups that create differences. The statistical significance level will be accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of rotator cuff tendinopathy,
* Having sufficient cooperation to perform the exercises.

Exclusion Criteria:

* Having a neurological problem,
* Having a previous fracture in the shoulder region,
* Having undergone a relevant surgery in the past,
* Having any chronic illness that could prevent exercise (e.g., chronic heart failure, pacemaker, etc.),
* Having a systemic condition that could affect proprioception, such as diabetes, rheumatoid arthritis, ankylosing spondylitis, or advanced osteoarthritis,
* Having received a physiotherapy program targeting the neck and upper extremity within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quick Disabilities of Arm, Shoulder & Hand | one day before the intervention and 6 weeks after
  The Quick Disabilities of Arm, Shoulder & Hand Index is used to measure upper extremity physical function. A Turkish validity and reliability study has been conducted. The scale includes 11 headings extracted from the long version. Each question consists of a 5-point scale. The total score is calculated with the formula [(sum of n responses) /n-1] ×25, where n= indicates the total number of questions answered. The total score varies between 0 (no disability) and 100 (severe disability). The final score is classified as; 0- 15: 'no problem', 16-40: 'problem but able to work', 40 and above: 'unable to work'.

SECONDARY OUTCOMES:
Shoulder Joint Range of Motion | one day before the intervention and 6 weeks after
  The range of motion of the shoulder joint will be measured in degrees using a standard goniometer. Measurements will be recorded for the shoulder joint in the directions of flexion, extension, abduction, adduction, internal rotation, and external rotation.
Assessment of Shoulder Pain | one day before the intervention and 6 weeks after
  The Visual Analog Scale (VAS) will be used to evaluate shoulder pain. Perceived pain ranges from no pain at all to extreme pain. According to the VAS, pain severity is rated as 'no pain' being 0 points and 'worst possible pain' being 10 points (on a 10 cm scale). The individual will be asked to mark the point on a 100-millimeter line that corresponds to their perceived pain level. The unit length from the point representing no pain to the individual's marked point indicates the level of pain. Pain levels are categorized as: <3 mild pain, 3-6 moderate pain, and >6 severe pain. Pain will be assessed in four different conditions: night pain, daytime pain, pain at rest, and pain during activity.
Western Ontario Rotator Cuff (WORC) Index | one day before the intervention and 6 weeks after
  The WORC is a self-assessment tool developed by Kirkley and colleagues in 2003 to measure the quality of life in individuals with rotator cuff tendinopathy. This scale consists of five subdomains: physical activities, sports/recreational activities, work, lifestyle, and emotions, and includes a total of 21 questions. The Turkish validity and reliability study has been conducted. The WORC index has been successfully translated and adapted into Turkish. The Turkish version of the WORC index is a reliable and valid tool for use in clinical studies with patients with rotator cuff tendinopathy.
Assessment of Hand Grip Strength: | one day before the intervention and 6 weeks after
  Hand grip strength is assessed using a dynamometer. In our study, a Jamar brand dynamometer will be used. The participant sits upright on an armless chair. Necessary precautions are taken to ensure the participant's posture remains stable during the measurement. The participant is instructed to grip the dynamometer as hard as possible while in shoulder adduction, elbow flexed at 90 degrees, and wrist in a mid-prone position. They are then told to release upon verbal command. The measurement is repeated three times separately, and the average value is recorded.
Assessment of Joint Position Sense: | one day before the intervention and 6 weeks after
  The joint position sense of the affected shoulder will be measured using a standard goniometer. The assessment will be done through an angle replication test, which evaluates the ability to actively replicate a predetermined angle. The specified angle is taught to the participant, and then they are asked to actively find the taught angle. The deviation between the angle found by the participant and the predetermined angle is recorded. The test will be performed in arm elevation positions including 30, 60, and 90 degrees of shoulder flexion and 30, 60, and 90 degrees of shoulder abduction. Each position will be repeated three times with the participant's eyes open, allowing them to memorize the position. After returning to the starting position, the participant's eyes will be closed, and they will be asked to repeat the same movement three times. After each movement, the goniometer will be positioned at the shoulder joint, and the physiotherapist will measure the angle.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Assist Prof, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhury S, Gwilym SE, Moser J, Carr AJ. Surgical options for patients with shoulder pain. Nat Rev Rheumatol. 2010 Apr;6(4):217-26. doi: 10.1038/nrrheum.2010.25. PMID 20357791
- [Background] Kibler WB. Rehabilitation of rotator cuff tendinopathy. Clin Sports Med. 2003 Oct;22(4):837-47. doi: 10.1016/s0278-5919(03)00048-6. PMID 14560550
- [Background] Arnocky SP, Lavagnino M, Egerbacher M. The Response of Tendon Cells to Changing Loads: Implications in the Etiopathogenesis of Tendinopathy. In: Woo L-Y, Renström AFH, Arnoczky SP, editors. Tendinopathy in athletes. Oxford, UK: Wiley online library; 2007. pp. 46-59.
- [Background] Camargo PR, Alburquerque-Sendin F, Salvini TF. Eccentric training as a new approach for rotator cuff tendinopathy: Review and perspectives. World J Orthop. 2014 Nov 18;5(5):634-44. doi: 10.5312/wjo.v5.i5.634. eCollection 2014 Nov 18. PMID 25405092
- [Background] Wulf G, Hoss M, Prinz W. Instructions for motor learning: differential effects of internal versus external focus of attention. J Mot Behav. 1998 Jun;30(2):169-79. doi: 10.1080/00222899809601334. PMID 20037032
- [Background] Wulf G, Lewthwaite R. Optimizing performance through intrinsic motivation and attention for learning: The OPTIMAL theory of motor learning. Psychon Bull Rev. 2016 Oct;23(5):1382-1414. doi: 10.3758/s13423-015-0999-9. PMID 26833314
- [Background] Wulf G, Weigelt M, Poulter D, McNevin N. Attentional focus on suprapostural tasks affects balance learning. Q J Exp Psychol A. 2003 Oct;56(7):1191-211. doi: 10.1080/02724980343000062. PMID 12959910
- [Background] Park SH, Yi CW, Shin JY, Ryu YU. Effects of external focus of attention on balance: a short review. J Phys Ther Sci. 2015 Dec;27(12):3929-31. doi: 10.1589/jpts.27.3929. Epub 2015 Dec 28. PMID 26834382
- [Background] Castillo-Vejar L, Lizama-Fuentes M, Bascour-Sandoval C, Cuyul-Vasquez I. [Attentional focus instructions for therapeutic exercise in people with musculoskeletal disorders. A scoping review]. Rehabilitacion (Madr). 2022 Oct-Dec;56(4):344-352. doi: 10.1016/j.rh.2021.11.006. Epub 2022 Apr 22. Spanish. PMID 35469643
- [Background] Lohse KR, Sherwood DE. Defining the focus of attention: effects of attention on perceived exertion and fatigue. Front Psychol. 2011 Nov 14;2:332. doi: 10.3389/fpsyg.2011.00332. eCollection 2011. PMID 22102843
- [Result] Hayes JR, Sheedy JE, Stelmack JA, Heaney CA. Computer use, symptoms, and quality of life. Optom Vis Sci. 2007 Aug;84(8):738-44. doi: 10.1097/OPX.0b013e31812f7546. PMID 17700327
- [Result] Bertelsen TI. [Visual coordination- and accommodation disturbances and eye diseases as causes of headache]. Nord Med. 1978 Apr;93(3-4):57-8. No abstract available. Norwegian. PMID 643521
- [Result] El O, Bircan C, Gulbahar S, Demiral Y, Sahin E, Baydar M, Kizil R, Griffin S, Akalin E. The reliability and validity of the Turkish version of the Western Ontario Rotator Cuff Index. Rheumatol Int. 2006 Oct;26(12):1101-8. doi: 10.1007/s00296-006-0151-2. Epub 2006 Jun 24. PMID 16799776
- [Result] Kirkley A, Alvarez C, Griffin S. The development and evaluation of a disease-specific quality-of-life questionnaire for disorders of the rotator cuff: The Western Ontario Rotator Cuff Index. Clin J Sport Med. 2003 Mar;13(2):84-92. doi: 10.1097/00042752-200303000-00004. PMID 12629425
- [Result] Koldas Dogan S, Ay S, Evcik D, Baser O. Adaptation of Turkish version of the questionnaire Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) in patients with carpal tunnel syndrome. Clin Rheumatol. 2011 Feb;30(2):185-91. doi: 10.1007/s10067-010-1470-y. Epub 2010 Apr 22. PMID 20411289
- [Result] Vafadar AK, Cote JN, Archambault PS. Interrater and Intrarater Reliability and Validity of 3 Measurement Methods for Shoulder-Position Sense. J Sport Rehabil. 2016 Feb 2;25(1):2014-0309. doi: 10.1123/jsr.2014-0309. Print 2016 Feb 1. PMID 25962861